CLINICAL TRIAL: NCT04560257
Title: Prone Positioning and High Flow Nasal Canula (HFNC) Therapy: A Game Changer in COVID-19 Outcome
Brief Title: High Flow Nasal Cannula HFNC In Covid-19 Patients
Acronym: HFNC19LGH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. M.Irfan Malik, Associate Professor of Pulmonology / Focal Person COVID-19, Lahore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH004
Record Dates: First submitted 2020-07-13; First posted 2020-09-23 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: SARS-CoV Infection; SARS (Severe Acute Respiratory Syndrome)
Keywords: COVID-19; High flow nasal cannula HFNC; Clinical outcome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: quasi- experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group intervene with HFNC (Experimental): Review effect of HFNC as clinical trial among hospitalized patients with COVID-19 infection.
  Interventions: Device: High flow nasal cannula HFNC

INTERVENTIONS:
Device: High flow nasal cannula HFNC — High flow nasal cannula HFNC is a device that delivered the warmed and humid air on high flow rate through nose. It is used to treat severe respiratory distress in COVID-19 patients, a non-invasive ventilatory approach which is relative comfortable by using humidified and pre-heated air containing large concentration of oxygen.
  Other Names: HFNC

SUMMARY:
Many non-invasive ventilatory choices are available for COVID-19 patient who are having mild to moderate respiratory distress and their use will decrease the chance of ICU admission, intubation and mechanical ventilation in severe cases of COVID-19. However, all these respiratory supports and oxygen supply devices are aerosol generating and their selection should be precised enough to control nosocomial spread.

High flow nasal cannula HFNC is a device that delivered the warmed and humid air on high flow rate through nose. It is used to treat severe respiratory distress in COVID-19 patients, a non-invasive ventilatory approach which is relative comfortable by using humidified and pre-heated air containing large concentration of oxygen. In acute respiratory failure HFNC is proven to be very effective and it also reduced the need of mechanical ventilation in severe patients. Apart from the supply of oxygen, HFNC generating positive airway pressure and decreasing the rebreathing from anatomical dead space.

Prone position is also a save therapy and has been proven to be effective for refractory hypoxia by increasing tidal volume, oxygenation and diaphragmatic functions in ARDS patients. Recent studies showed that prone positioning and HFNC might avoid the prerequisite of intubation in moderate to severe patients of ARDS and as a result it decreases the nosocomial infection in physicians who are doing these aerosol generating procedures.

DETAILED DESCRIPTION:
This is observational single-center study, that will be done at Lahore General Hospital in which 95 beds are allocated for COVID-19 patients including ICUs and HDUs. Ethical approval will be obtained from research ethical committee of Lahore General hospital, Lahore. Informed consent will be obtained from all patients who will agree to publish their data in this research. We will protect patient's privacy and obey with the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* All patients of > 18 years of ages, males and females who will be diagnosed COVID-19 positive by RT-PCR with moderate illness.
* Patients having classical radiological lesions of COVID-19 on X-ray chest or HRCT chest.
* Respiratory rate > 30/ min and not responding to non-rebreather masks.
* COVID-related pneumonia requiring non-invasive ventilatory support (high-flow nasal cannula, and / or non-invasive ventilation and / or CPAP)

Exclusion Criteria:

* Inability to provide consent;
* Severe respiratory failure requiring invasive ventilatory support;
* Indication of immediate tracheal intubation
* Significant acute progressive circulatory insufficiency
* Impaired alertness, confusion, restlessness
* Chest trauma or other contraindication to prone position
* Pneumothorax
* Nasal blockade
* Unable to tolerate high flow oxygen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response of HFNC | 10 days
  The number of patients treated with non-invasive ventilation devices. HFNC related events (hot air feeling, nasal lesions)

SECONDARY OUTCOMES:
Duration of intervention | 15 days
  Length of HFNC therapy to COVID-19 patients
Duration of hospitalization | 15 days
  Number of days of hospital admission either in ICU or HDUs till date of discharge
Supplemental Oxygen Requirement from Baseline | 15 days
  Duration of increased supplemental oxygen requirement from baseline
Radiological outcome | 15 days
  Follow up radiological response HR-CT.

CONTACTS AND LOCATIONS:
Overall Officials: Sardar Al-Fareed Zafar, Study Director — Post-Graduate Medical Institute, Lahore General Hospital, Lahore Pakistan
Locations (1):
- Muhammad Irfan Malik, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whittle JS, Pavlov I, Sacchetti AD, Atwood C, Rosenberg MS. Respiratory support for adult patients with COVID-19. J Am Coll Emerg Physicians Open. 2020 Apr 13;1(2):95-101. doi: 10.1002/emp2.12071. eCollection 2020 Apr. PMID 32427171
- [Background] Richards M, Le Roux D, Cooke L, Argent A. The Influence of High Flow Nasal Cannulae on the Outcomes of Severe Respiratory Disease in Children Admitted to a Regional Hospital in South Africa. J Trop Pediatr. 2020 Dec 1;66(6):612-620. doi: 10.1093/tropej/fmaa024. PMID 32533147
- [Background] Pinkham M, Tatkov S. Effect of flow and cannula size on generated pressure during nasal high flow. Crit Care. 2020 May 24;24(1):248. doi: 10.1186/s13054-020-02980-w. No abstract available. PMID 32448344
- [Background] Tu GW, Liao YX, Li QY, Dong H, Yang LY, Zhang XY, Fu SZ, Wang RL. Prone positioning in high-flow nasal cannula for COVID-19 patients with severe hypoxemia: a pilot study. Ann Transl Med. 2020 May;8(9):598. doi: 10.21037/atm-20-3005. No abstract available. PMID 32566624